CLINICAL TRIAL: NCT00593450
Title: Comparison of Age-related Macular Degeneration Treatments Trials: Lucentis-Avastin Trial (CATT)
Brief Title: Comparison of Age-related Macular Degeneration Treatments Trials: Lucentis-Avastin Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEI-137; U10EY017823 (NIH)
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Age Related Macular Degeneration
Keywords: bevacizumab; ranibizumab; choroidal neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1 (Active Comparator): Lucentis® on a fixed schedule of every 4 weeks for 1 year; at 1 year, re-randomization to Lucentis® every 4 weeks or to variable dosing.
  Interventions: Drug: ranibizumab
- 2 (Experimental): Avastin® on a fixed schedule of every 4 weeks for 1 year; at 1 year, re-randomization to Avastin® every 4 weeks or to variable dosing.
  Interventions: Drug: bevacizumab
- 3 (Experimental): Lucentis® on a variable dosing schedule for 2 years; i.e., after initial treatment, monthly evaluation for treatment based on signs of lesion activity.
  Interventions: Drug: ranibizumab
- 4 (Experimental): Avastin® on a variable dosing schedule for 2 years; i.e., after initial treatment, monthly evaluation for treatment based on signs of lesion activity.
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: ranibizumab — • 0.5 mg (0.05 mL)intravitreal injection
  Other Names: Lucentis
  Arms: 1; 3
Drug: bevacizumab — • 1.25 mg (0.05 mL)intravitreal injection
  Other Names: Avastin
  Arms: 2; 4

SUMMARY:
The purpose of the study is to evaluate the relative efficacy and safety of treatment of neovascular AMD with Lucentis on a fixed schedule, Avastin on a fixed schedule, Lucentis on a variable schedule, and Avastin on a variable schedule.

A five year follow-up visit is being conducted in 2014 to gather information on long term outcomes.

DETAILED DESCRIPTION:
Age related macular degeneration (AMD) is the leading cause of severe vision loss in people over the age of 65 in the United States and other Western countries. More than 1.6 million people in the US currently have one or both eyes affected by the advanced stage of AMD.

Lucentis® is the most effective treatment for neovascular AMD studied to date. Bevacizumab (Avastin®) and Lucentis® are derived from the same monoclonal antibody. Following the encouraging clinical trial results with Lucentis®, several investigators began evaluating intravitreal Avastin® for the treatment of CNV. Given its molecular similarity to Lucentis, its low cost, and its availability, the interest in Avastin® has been considerable. Avastin® has not been evaluated relative to Lucentis®.

In addition, previous studies do not answer the question of whether a reduced dosing schedule is as effective as a fixed schedule of monthly injections. Treatment dependent on clinical response has the potential to reduce the treatment burden to patients as well as to reduce the overall cost of therapy.

Only a single eye in each patient was analyzed.

At the five year follow-up visit, the subjects will undergo the same examinations and procedures as in the original study; however, the five year follow-up visit deos not involve any study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Active, subfoveal choroidal neovascularization (CNV)
* Fibrosis < 50% of total lesion area
* Visual acuity (VA) 20/25-20/320
* Age ≥ 50 yrs
* At least 1 drusen (>63μ) in either eye or late AMD in fellow eye

Exclusion Criteria:

* Previous treatment for CNV in study eye
* Other progressive retinal disease likely to compromise VA
* Contraindications to injections with Lucentis or Avastin

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1208 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Martin, MD, Study Chair — The Cleveland Clinic; Stuart L Fine, MD, Study Chair — Study Vice-Chair, University of Pennsylvania; Maureen G Maguire, PhD, Study Director — Director of Coordinating Center, University of Pennsylvania; Glenn Jaffe,, MD, Study Director — Director of OCT Reading Center, Duke University; Juan E Grunwald, MD, Principal Investigator — Principal Investigator of Photography Reading Center, Universisty of Pennsylvania
Locations (58):
- United States (58):
  - Retina Consultants of Arizona, Mesa, Arizona
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Retina Associates Southwest, P.C., Tucson, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - University of California-Davis Medical Center, Sacramento, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - West Coast Retina Medical Group, Inc., San Francisco, California
  - California Retinal Consultants, Santa Barbara, California
  - West Coast Retina Medical Group, Inc., Walnut Creek, California
  - Colorado Retina Associates, Denver, Colorado
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Illinois Retina Associates, Flossmoor, Illinois
  - Ingalls Memorial Hospital/Illinois Retina Associates, Harvey, Illinois
  - Illinois Retina Associates, Joliet, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Retina Associates of Kentucky, Lexington, Kentucky
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Elman Retina Group, P.A., Baltimore, Maryland
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Retina Specialists, Towson, Maryland
  - Massachusetts Eye & Ear Infirmary, Boston, Massachusetts
  - Opthalmic Consultants of Boston, Boston, Massachusetts
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Vision Research Foundation/Associated Retinal Consultants, P.C., Grand Rapids, Michigan
  - Vision Research Foundation/Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - Vision research Foundation/Associated Retinal Consultants. P.C., Traverse City, Michigan
  - VitreoRetinal Surgery, Edina, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Barnes Retina Institute, St Louis, Missouri
  - Retina Vitreous Center, PA, New Brunswick, New Jersey
  - Retina Vitreous Center, PA, Toms River, New Jersey
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - Long Island Vitreoretinal Consultants, Riverhead, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, nose & Throat Associates, Charlotte, North Carolina
  - Duke University Eye Center, Durham, North Carolina
  - Charlotte Eye,Ear, Nose & Throat Associates, Monroe, North Carolina
  - Retina Associates of Cleveland, Beachwood, Ohio
  - Ohio State University Eye Physicians & Surgeons-Retina Division, Dublin, Ohio
  - Retina Associates of Cleveland, Inc., Lakewood, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Northwest, P.C., Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Retina Diagnostic and Treatment Associates, LLC, Philadelphia, Pennsylvania
  - Retina Vitreous Consultants, Pittsburgh, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Retina Vitreous Associates, P.C., Nashville, Tennessee
  - Texas Retina Associates, Arlington, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - The Retina Group of Washington, Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Available at https://hyperprod.cceb.med.upenn.edu/catt/catt_index.php

REFERENCES:
- [Background] Martin DF, Maguire MG, Fine SL. Identifying and eliminating the roadblocks to comparative-effectiveness research. N Engl J Med. 2010 Jul 8;363(2):105-7. doi: 10.1056/NEJMp1001201. Epub 2010 Jun 2. No abstract available. PMID 20519677
- [Result] CATT Research Group; Martin DF, Maguire MG, Ying GS, Grunwald JE, Fine SL, Jaffe GJ. Ranibizumab and bevacizumab for neovascular age-related macular degeneration. N Engl J Med. 2011 May 19;364(20):1897-908. doi: 10.1056/NEJMoa1102673. Epub 2011 Apr 28. PMID 21526923
- [Result] Comparison of Age-related Macular Degeneration Treatments Trials (CATT) Research Group; Martin DF, Maguire MG, Fine SL, Ying GS, Jaffe GJ, Grunwald JE, Toth C, Redford M, Ferris FL 3rd. Ranibizumab and bevacizumab for treatment of neovascular age-related macular degeneration: two-year results. Ophthalmology. 2012 Jul;119(7):1388-98. doi: 10.1016/j.ophtha.2012.03.053. Epub 2012 May 1. PMID 22555112
- [Result] Grunwald JE, Daniel E, Ying GS, Pistilli M, Maguire MG, Alexander J, Whittock-Martin R, Parker CR, Sepielli K, Blodi BA, Martin DF; CATT Research Group. Photographic assessment of baseline fundus morphologic features in the Comparison of Age-Related Macular Degeneration Treatments Trials. Ophthalmology. 2012 Aug;119(8):1634-41. doi: 10.1016/j.ophtha.2012.02.013. Epub 2012 Apr 17. PMID 22512984
- [Result] Martin DF, Maguire MG, Fine SL. Bevacizumab: not as good with more adverse reactions? Response. Clin Exp Ophthalmol. 2011 Sep-Oct;39(7):718-20. doi: 10.1111/j.1442-9071.2011.02703.x. No abstract available. PMID 22452699
- [Result] Cheung CM, Wong TY. Ranibizumab and bevacizumab for AMD. N Engl J Med. 2011 Dec 8;365(23):2237; author reply 2237. doi: 10.1056/NEJMc1107895. No abstract available. PMID 22150050
- [Result] DeCroos FC, Toth CA, Stinnett SS, Heydary CS, Burns R, Jaffe GJ; CATT Research Group. Optical coherence tomography grading reproducibility during the Comparison of Age-related Macular Degeneration Treatments Trials. Ophthalmology. 2012 Dec;119(12):2549-57. doi: 10.1016/j.ophtha.2012.06.040. Epub 2012 Aug 28. PMID 22939114
- [Result] Ying GS, Huang J, Maguire MG, Jaffe GJ, Grunwald JE, Toth C, Daniel E, Klein M, Pieramici D, Wells J, Martin DF; Comparison of Age-related Macular Degeneration Treatments Trials Research Group. Baseline predictors for one-year visual outcomes with ranibizumab or bevacizumab for neovascular age-related macular degeneration. Ophthalmology. 2013 Jan;120(1):122-9. doi: 10.1016/j.ophtha.2012.07.042. Epub 2012 Oct 6. PMID 23047002
- [Result] Hagstrom SA, Ying GS, Pauer GJT, Sturgill-Short GM, Huang J, Callanan DG, Kim IK, Klein ML, Maguire MG, Martin DF; Comparison of AMD Treatments Trials Research Group. Pharmacogenetics for genes associated with age-related macular degeneration in the Comparison of AMD Treatments Trials (CATT). Ophthalmology. 2013 Mar;120(3):593-599. doi: 10.1016/j.ophtha.2012.11.037. Epub 2013 Jan 18. PMID 23337555
- [Result] Jaffe GJ, Martin DF, Toth CA, Daniel E, Maguire MG, Ying GS, Grunwald JE, Huang J; Comparison of Age-related Macular Degeneration Treatments Trials Research Group. Macular morphology and visual acuity in the comparison of age-related macular degeneration treatments trials. Ophthalmology. 2013 Sep;120(9):1860-70. doi: 10.1016/j.ophtha.2013.01.073. Epub 2013 May 1. PMID 23642377
- [Result] Maguire MG, Daniel E, Shah AR, Grunwald JE, Hagstrom SA, Avery RL, Huang J, Martin RW, Roth DB, Castellarin AA, Bakri SJ, Fine SL, Martin DF; Comparison of Age-Related Macular Degeneration Treatments Trials (CATT Research Group). Incidence of choroidal neovascularization in the fellow eye in the comparison of age-related macular degeneration treatments trials. Ophthalmology. 2013 Oct;120(10):2035-41. doi: 10.1016/j.ophtha.2013.03.017. Epub 2013 May 22. PMID 23706946
- [Result] Daniel E, Toth CA, Grunwald JE, Jaffe GJ, Martin DF, Fine SL, Huang J, Ying GS, Hagstrom SA, Winter K, Maguire MG; Comparison of Age-related Macular Degeneration Treatments Trials Research Group. Risk of scar in the comparison of age-related macular degeneration treatments trials. Ophthalmology. 2014 Mar;121(3):656-66. doi: 10.1016/j.ophtha.2013.10.019. Epub 2013 Dec 4. PMID 24314839
- [Result] Grunwald JE, Daniel E, Huang J, Ying GS, Maguire MG, Toth CA, Jaffe GJ, Fine SL, Blodi B, Klein ML, Martin AA, Hagstrom SA, Martin DF; CATT Research Group. Risk of geographic atrophy in the comparison of age-related macular degeneration treatments trials. Ophthalmology. 2014 Jan;121(1):150-161. doi: 10.1016/j.ophtha.2013.08.015. Epub 2013 Sep 29. PMID 24084496
- [Result] Hagstrom SA, Ying GS, Pauer GJ, Sturgill-Short GM, Huang J, Maguire MG, Martin DF; Comparison of Age-Related Macular Degeneration Treatments Trials (CATT) Research Group. VEGFA and VEGFR2 gene polymorphisms and response to anti-vascular endothelial growth factor therapy: comparison of age-related macular degeneration treatments trials (CATT). JAMA Ophthalmol. 2014 May;132(5):521-7. doi: 10.1001/jamaophthalmol.2014.109. PMID 24652518
- [Result] Kim BJ, Ying GS, Huang J, Levy NE, Maguire MG; CATT Research Group. Sporadic visual acuity loss in the Comparison of Age-Related Macular Degeneration Treatments Trials (CATT). Am J Ophthalmol. 2014 Jul;158(1):128-135.e10. doi: 10.1016/j.ajo.2014.04.004. Epub 2014 Apr 13. PMID 24727261
- [Result] Folgar FA, Jaffe GJ, Ying GS, Maguire MG, Toth CA; Comparison of Age-Related Macular Degeneration Treatments Trials Research Group. Comparison of optical coherence tomography assessments in the comparison of age-related macular degeneration treatments trials. Ophthalmology. 2014 Oct;121(10):1956-65. doi: 10.1016/j.ophtha.2014.04.020. Epub 2014 May 15. PMID 24835760
- [Result] Ying GS, Kim BJ, Maguire MG, Huang J, Daniel E, Jaffe GJ, Grunwald JE, Blinder KJ, Flaxel CJ, Rahhal F, Regillo C, Martin DF; CATT Research Group. Sustained visual acuity loss in the comparison of age-related macular degeneration treatments trials. JAMA Ophthalmol. 2014 Aug;132(8):915-21. doi: 10.1001/jamaophthalmol.2014.1019. PMID 24875610
- [Result] Gewaily DY, Grunwald JE, Pistilli M, Ying GS, Maguire MG, Daniel E, Ostroff CP, Fine SL; CATT Research Group. Delayed patchy choroidal filling in the Comparison of Age-Related Macular Degeneration Treatments Trials (CATT). Am J Ophthalmol. 2014 Sep;158(3):525-31.e2. doi: 10.1016/j.ajo.2014.06.004. Epub 2014 Jun 17. PMID 24949820
- [Result] Lee JY, Folgar FA, Maguire MG, Ying GS, Toth CA, Martin DF, Jaffe GJ; CATT Research Group. Outer retinal tubulation in the comparison of age-related macular degeneration treatments trials (CATT). Ophthalmology. 2014 Dec;121(12):2423-31. doi: 10.1016/j.ophtha.2014.06.013. Epub 2014 Jul 23. PMID 25064723
- [Result] Moja L, Lucenteforte E, Kwag KH, Bertele V, Campomori A, Chakravarthy U, D'Amico R, Dickersin K, Kodjikian L, Lindsley K, Loke Y, Maguire M, Martin DF, Mugelli A, Muhlbauer B, Puntmann I, Reeves B, Rogers C, Schmucker C, Subramanian ML, Virgili G. Systemic safety of bevacizumab versus ranibizumab for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2014 Sep 15;9(9):CD011230. doi: 10.1002/14651858.CD011230.pub2. PMID 25220133
- [Result] Altaweel MM, Daniel E, Martin DF, Mittra RA, Grunwald JE, Lai MM, Melamud A, Morse LS, Huang J, Ferris FL 3rd, Fine SL, Maguire MG; Comparison of Age-related Macular Degeneration Treatments Trials (CATT) Research Group; Comparison of Age-related Macular Degeneration Treatments Trials CATT Research Group. Outcomes of eyes with lesions composed of >50% blood in the Comparison of Age-related Macular Degeneration Treatments Trials (CATT). Ophthalmology. 2015 Feb;122(2):391-398.e5. doi: 10.1016/j.ophtha.2014.08.020. Epub 2014 Oct 11. PMID 25307130
- [Result] Grunwald JE, Pistilli M, Ying GS, Maguire MG, Daniel E, Martin DF; Comparison of Age-related Macular Degeneration Treatments Trials Research Group. Growth of geographic atrophy in the comparison of age-related macular degeneration treatments trials. Ophthalmology. 2015 Apr;122(4):809-16. doi: 10.1016/j.ophtha.2014.11.007. Epub 2014 Dec 24. PMID 25542520
- [Result] Meredith TA, McCannel CA, Barr C, Doft BH, Peskin E, Maguire MG, Martin DF, Prenner JL; Comparison of Age-Related Macular Degeneration Treatments Trials Research Group. Postinjection endophthalmitis in the comparison of age-related macular degeneration treatments trials (CATT). Ophthalmology. 2015 Apr;122(4):817-21. doi: 10.1016/j.ophtha.2014.10.027. Epub 2015 Jan 15. PMID 25600198
- [Result] Toth CA, Decroos FC, Ying GS, Stinnett SS, Heydary CS, Burns R, Maguire M, Martin D, Jaffe GJ. IDENTIFICATION OF FLUID ON OPTICAL COHERENCE TOMOGRAPHY BY TREATING OPHTHALMOLOGISTS VERSUS A READING CENTER IN THE COMPARISON OF AGE-RELATED MACULAR DEGENERATION TREATMENTS TRIALS. Retina. 2015 Jul;35(7):1303-14. doi: 10.1097/IAE.0000000000000483. PMID 26102433
- [Result] Ciulla TA, Ying GS, Maguire MG, Martin DF, Jaffe GJ, Grunwald JE, Daniel E, Toth CA; Comparison of Age-Related Macular Degeneration Treatments Trials Research Group. Influence of the Vitreomacular Interface on Treatment Outcomes in the Comparison of Age-Related Macular Degeneration Treatments Trials. Ophthalmology. 2015 Jun;122(6):1203-11. doi: 10.1016/j.ophtha.2015.02.031. Epub 2015 Mar 29. PMID 25824327
- [Result] Hagstrom SA, Ying GS, Maguire MG, Martin DF; CATT Research Group; Gibson J, Lotery A, Chakravarthy U; IVAN Study Investigators. VEGFR2 Gene Polymorphisms and Response to Anti-Vascular Endothelial Growth Factor Therapy in Age-Related Macular Degeneration. Ophthalmology. 2015 Aug;122(8):1563-8. doi: 10.1016/j.ophtha.2015.04.024. Epub 2015 May 28. PMID 26028346
- [Result] Willoughby AS, Ying GS, Toth CA, Maguire MG, Burns RE, Grunwald JE, Daniel E, Jaffe GJ; Comparison of Age-Related Macular Degeneration Treatments Trials Research Group. Subretinal Hyperreflective Material in the Comparison of Age-Related Macular Degeneration Treatments Trials. Ophthalmology. 2015 Sep;122(9):1846-53.e5. doi: 10.1016/j.ophtha.2015.05.042. Epub 2015 Jul 2. PMID 26143666
- [Result] Ying GS, Maguire MG, Daniel E, Ferris FL, Jaffe GJ, Grunwald JE, Toth CA, Huang J, Martin DF; Comparison of Age-Related Macular Degeneration Treatments Trials (CATT) Research Group. Association of Baseline Characteristics and Early Vision Response with 2-Year Vision Outcomes in the Comparison of AMD Treatments Trials (CATT). Ophthalmology. 2015 Dec;122(12):2523-31.e1. doi: 10.1016/j.ophtha.2015.08.015. Epub 2015 Sep 15. PMID 26383996
- [Result] Ying GS, Maguire MG, Daniel E, Grunwald JE, Ahmed O, Martin DF; Comparison of Age-Related Macular Degeneration Treatments Trials Research Group. Association between Antiplatelet or Anticoagulant Drugs and Retinal or Subretinal Hemorrhage in the Comparison of Age-Related Macular Degeneration Treatments Trials. Ophthalmology. 2016 Feb;123(2):352-360. doi: 10.1016/j.ophtha.2015.09.046. Epub 2015 Nov 4. PMID 26545320
- [Result] Daniel E, Shaffer J, Ying GS, Grunwald JE, Martin DF, Jaffe GJ, Maguire MG; Comparison of Age-Related Macular Degeneration Treatments Trials (CATT) Research Group. Outcomes in Eyes with Retinal Angiomatous Proliferation in the Comparison of Age-Related Macular Degeneration Treatments Trials (CATT). Ophthalmology. 2016 Mar;123(3):609-16. doi: 10.1016/j.ophtha.2015.10.034. Epub 2015 Dec 8. PMID 26681392
- [Result] Shah N, Maguire MG, Martin DF, Shaffer J, Ying GS, Grunwald JE, Toth CA, Jaffe GJ, Daniel E; Comparison of Age-related Macular Degeneration Treatments Trials Research Group. Angiographic Cystoid Macular Edema and Outcomes in the Comparison of Age-Related Macular Degeneration Treatments Trials. Ophthalmology. 2016 Apr;123(4):858-64. doi: 10.1016/j.ophtha.2015.11.030. Epub 2016 Jan 8. PMID 26778329
- [Result] Sharma S, Toth CA, Daniel E, Grunwald JE, Maguire MG, Ying GS, Huang J, Martin DF, Jaffe GJ; Comparison of Age-related Macular Degeneration Treatments Trials Research Group. Macular Morphology and Visual Acuity in the Second Year of the Comparison of Age-Related Macular Degeneration Treatments Trials. Ophthalmology. 2016 Apr;123(4):865-75. doi: 10.1016/j.ophtha.2015.12.002. Epub 2016 Jan 9. PMID 26783095
- [Result] Zhou Q, Daniel E, Maguire MG, Grunwald JE, Martin ER, Martin DF, Ying GS; Comparison of Age-Related Macular Degeneration Treatments Trials Research Group. Pseudodrusen and Incidence of Late Age-Related Macular Degeneration in Fellow Eyes in the Comparison of Age-Related Macular Degeneration Treatments Trials. Ophthalmology. 2016 Jul;123(7):1530-40. doi: 10.1016/j.ophtha.2016.02.043. Epub 2016 Apr 1. PMID 27040149
- [Result] Maguire MG, Ying GS, Jaffe GJ, Toth CA, Daniel E, Grunwald J, Martin DF, Hagstrom SA; CATT Research Group. Single-Nucleotide Polymorphisms Associated With Age-Related Macular Degeneration and Lesion Phenotypes in the Comparison of Age-Related Macular Degeneration Treatments Trials. JAMA Ophthalmol. 2016 Jun 1;134(6):674-81. doi: 10.1001/jamaophthalmol.2016.0669. PMID 27099955
- [Derived] Core JQ, Hua P, Daniel E, Grunwald JE, Jaffe G, Maguire MG, Ying GS; Comparison of Age-related Macular Degeneration Treatments Trials (CATT) Research Group. Thiazolidinedione use and retinal fluid in the comparison of age-related macular degeneration treatments trials. Br J Ophthalmol. 2023 Jul;107(7):1000-1006. doi: 10.1136/bjophthalmol-2021-320665. Epub 2022 Apr 15. PMID 35428655
- [Derived] Core JQ, Pistilli M, Hua P, Daniel E, Grunwald JE, Toth CA, Jaffe GJ, Martin DF, Maguire MG, Ying GS; Comparison of Age-related Macular Degeneration Treatments Trials (CATT) Research Group. Predominantly Persistent Intraretinal Fluid in the Comparison of Age-related Macular Degeneration Treatments Trials. Ophthalmol Retina. 2022 Sep;6(9):771-785. doi: 10.1016/j.oret.2022.03.024. Epub 2022 Apr 9. PMID 35405352
- [Derived] Kolomeyer AM, Smith E, Daniel E, Ying GS, Pan W, Pistilli M, Grunwald J, Maguire MG, Kim BJ; CATT Research Group. BETA-PERIPAPILLARY ATROPHY AND GEOGRAPHIC ATROPHY IN THE COMPARISON OF AGE-RELATED MACULAR DEGENERATION TREATMENTS TRIALS. Retina. 2021 Jan 1;41(1):125-134. doi: 10.1097/IAE.0000000000002825. PMID 32383840
- [Derived] Li E, Donati S, Lindsley KB, Krzystolik MG, Virgili G. Treatment regimens for administration of anti-vascular endothelial growth factor agents for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 May 5;5(5):CD012208. doi: 10.1002/14651858.CD012208.pub2. PMID 32374423
- [Derived] Daniel E, Maguire MG, Grunwald JE, Toth CA, Jaffe GJ, Martin DF, Ying GS; Comparison of Age-Related Macular Degeneration Treatments Trials Research Group. Incidence and Progression of Nongeographic Atrophy in the Comparison of Age-Related Macular Degeneration Treatments Trials (CATT) Clinical Trial. JAMA Ophthalmol. 2020 May 1;138(5):510-518. doi: 10.1001/jamaophthalmol.2020.0437. PMID 32191267
- [Derived] Ramakrishnan MS, Yu Y, VanderBeek BL. Association of Visit Adherence and Visual Acuity in Patients With Neovascular Age-Related Macular Degeneration: Secondary Analysis of the Comparison of Age-Related Macular Degeneration Treatment Trial. JAMA Ophthalmol. 2020 Mar 1;138(3):237-242. doi: 10.1001/jamaophthalmol.2019.4577. PMID 32027349
- [Derived] Scoles D, Ying GS, Pan W, Hua P, Grunwald JE, Daniel E, Jaffe GJ, Toth CA, Martin DF, Maguire MG; Comparison of AMD Treatments Trials Research Group. Characteristics of Eyes With Good Visual Acuity at 5 Years After Initiation of Treatment for Age-Related Macular Degeneration but Not Receiving Treatment From Years 3 to 5: Post Hoc Analysis of the CATT Randomized Clinical Trial. JAMA Ophthalmol. 2020 Mar 1;138(3):276-284. doi: 10.1001/jamaophthalmol.2019.5831. PMID 31999297
- [Derived] Bavinger JC, Ying GS, Daniel E, Grunwald JE, Maguire MG; Comparison of Age-Related Macular Degeneration Treatments Trials Research Group. Association Between Cilioretinal Arteries and Advanced Age-Related Macular Degeneration: Secondary Analysis of the Comparison of Age-Related Macular Degeneration Treatment Trials (CATT). JAMA Ophthalmol. 2019 Nov 1;137(11):1306-1311. doi: 10.1001/jamaophthalmol.2019.3509. PMID 31513262
- [Derived] Toth CA, Tai V, Pistilli M, Chiu SJ, Winter KP, Daniel E, Grunwald JE, Jaffe GJ, Martin DF, Ying GS, Farsiu S, Maguire MG; Comparison of Age-related Macular Degeneration Treatments Trials Research Group. Distribution of OCT Features within Areas of Macular Atrophy or Scar after 2 Years of Anti-VEGF Treatment for Neovascular AMD in CATT. Ophthalmol Retina. 2019 Apr;3(4):316-325. doi: 10.1016/j.oret.2018.11.011. Epub 2018 Dec 3. PMID 31014683
- [Derived] Daniel E, Ying GS, Kim BJ, Toth CA, Ferris F 3rd, Martin DF, Grunwald JE, Jaffe GJ, Dunaief JL, Pan W, Maguire MG; Comparison of Age-Related Macular Degeneration Treatments Trials. Five-Year Follow-up of Nonfibrotic Scars in the Comparison of Age-Related Macular Degeneration Treatments Trials. Ophthalmology. 2019 May;126(5):743-751. doi: 10.1016/j.ophtha.2018.11.020. Epub 2018 Nov 23. PMID 30476517
- [Derived] Jaffe GJ, Ying GS, Toth CA, Daniel E, Grunwald JE, Martin DF, Maguire MG; Comparison of Age-related Macular Degeneration Treatments Trials Research Group. Macular Morphology and Visual Acuity in Year Five of the Comparison of Age-related Macular Degeneration Treatments Trials. Ophthalmology. 2019 Feb;126(2):252-260. doi: 10.1016/j.ophtha.2018.08.035. Epub 2018 Sep 3. PMID 30189282
- [Derived] Daniel E, Pan W, Ying GS, Kim BJ, Grunwald JE, Ferris FL 3rd, Jaffe GJ, Toth CA, Martin DF, Fine SL, Maguire MG; Comparison of Age-related Macular Degeneration Treatments Trials. Development and Course of Scars in the Comparison of Age-Related Macular Degeneration Treatments Trials. Ophthalmology. 2018 Jul;125(7):1037-1046. doi: 10.1016/j.ophtha.2018.01.004. Epub 2018 Feb 14. PMID 29454660
- [Derived] Grunwald JE, Pistilli M, Daniel E, Ying GS, Pan W, Jaffe GJ, Toth CA, Hagstrom SA, Maguire MG, Martin DF; Comparison of Age-Related Macular Degeneration Treatments Trials Research Group. Incidence and Growth of Geographic Atrophy during 5 Years of Comparison of Age-Related Macular Degeneration Treatments Trials. Ophthalmology. 2017 Jan;124(1):97-104. doi: 10.1016/j.ophtha.2016.09.012. Epub 2016 Oct 27. PMID 28079023
- See also: Click here for more information about this study: Comparison of AMD Treatments Trials (CATT) — http://www.med.upenn.edu/cpob/catt.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note: The Data and Safety Monitoring Committee for CATT recommended excluding the data for all patients (N=23) from one center because of serious protocol non-compliance. Unless specified otherwise, only the 1185 patients enrolled by the remaining 43 centers are included in analyses.
Groups:
- 1-Lucentis Monthly: Lucentis® on a fixed schedule of every 4 weeks for 1 year; at 1 year, re-randomization to Lucentis® every 4 weeks or to variable dosing.
- 2-Avastin Monthly: Avastin® on a fixed schedule of every 4 weeks for 1 year; at 1 year, re-randomization to Avastin® every 4 weeks or to variable dosing.
- 3-Lucentis as Needed: Lucentis® on a variable dosing schedule for 2 years; i.e., after initial treatment, monthly evaluation for treatment based on signs of lesion activity.
- 4-Avastin as Needed: Avastin® on a variable dosing schedule for 2 years; i.e., after initial treatment, monthly evaluation for treatment based on signs of lesion activity.
Period: Overall Study
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Started | 301 | 286 | 298 | 300
Completed | 284 | 265 | 285 | 271
Not Completed | 17 | 21 | 13 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed | Total
Number analyzed (Participants) | 301 | 286 | 298 | 300 | 1185
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (7.4) | 80.1 (7.3) | 78.4 (7.8) | 79.3 (7.6) | 79.3 (7.5)
Age, Customized [Number; unit: participants]
  50-59 years | 2 | 1 | 6 | 2 | 11
  60-69 years | 33 | 28 | 31 | 34 | 126
  70-79 years | 102 | 84 | 115 | 103 | 404
  80-89 years | 142 | 150 | 126 | 142 | 560
  >=90 years | 22 | 23 | 20 | 19 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 180 | 185 | 184 | 732
  Male | 118 | 106 | 113 | 116 | 453
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 297 | 281 | 296 | 294 | 1168
  Other | 4 | 5 | 2 | 6 | 17
History of myocardial infarction [Number; unit: Participants]
  Yes | 34 | 40 | 30 | 36 | 140
  No | 267 | 246 | 268 | 264 | 1045
History of stroke [Number; unit: Participants]
  Yes | 14 | 18 | 22 | 16 | 70
  No | 287 | 268 | 276 | 284 | 1115
History of transient ischemic attack [Number; unit: Participants]
  Yes | 12 | 25 | 12 | 19 | 68
  No | 289 | 261 | 286 | 281 | 1117
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 134 (18) | 135 (19) | 136 (17) | 135 (17) | 135 (18)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 75 (10) | 75 (10) | 76 (9) | 75 (10) | 75 (10)
Visual-acuity score and Snellen equivalent [Number; unit: Participants]
  68-82 letters, 20/25-40 | 111 | 94 | 116 | 103 | 424
  53-67 letters, 20/50-80 | 98 | 118 | 108 | 119 | 443
  38-52 letters, 20/100-160 | 67 | 53 | 58 | 58 | 236
  23-37 letters, 20/200-320 | 25 | 21 | 16 | 20 | 82
Visual-acuity score and Snellen equivalent [Mean (Standard Deviation); unit: Letters] — Visual acuity testing was performed with the Electronic Visual Tester (EVA) following the ETDRS protocol. VA score is measured as number of letters read correctly.
  In this study, the visual acuity letter score is ranged from 23 to 82, with the higher score the better visual acuity.
  Letters | 60.1 (14.3) | 60.2 (13.1) | 61.5 (13.2) | 60.4 (13.4) | 60.5 (13.5)
Total thickness at fovea [Mean (Standard Deviation); unit: μm] | 458 (184) | 463 (196) | 458 (193) | 461 (175) | 460 (187)
Retinal thickness plus subfoveal-fluid thickness at fovea [Mean (Standard Deviation); unit: microns] | 251 (122) | 254 (121) | 247 (122) | 252 (115) | 251 (120)
Foveal center involvement [Number; unit: Participants]
  Choroidal neovacularization | 176 | 153 | 176 | 183 | 688
  Fluid | 85 | 81 | 77 | 72 | 315
  Hemorrhage | 20 | 24 | 24 | 25 | 93
  Other | 18 | 20 | 15 | 18 | 71
  No choroidal neovascularization or can't grade | 2 | 8 | 6 | 2 | 18

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline Visual-acuity Score (Frequency)
Time Frame: Baseline and 1 Year
Measure: Number; unit: Participants
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 284 | 265 | 285 | 271
Participants
  Increase of ≥15 letters | 97 | 83 | 71 | 76
  Increase of 5-14 letters | 90 | 98 | 103 | 90
  Change of ≤4 letters | 62 | 50 | 75 | 59
  Decrease of 5-14 letters | 19 | 18 | 23 | 23
  Decrease of ≥15 letters | 16 | 16 | 13 | 23

2. Primary Outcome: Change From Baseline in Visual-acuity Score (Continuous)
Description: Visual acuity testing was performed with the Electronic Visual Tester (EVA) following the ETDRS protocol. VA score is measured as number of letters read correctly. The VA score change is the difference of the VA score at 1 Year and the VA score at baseline.
  In this study, the outcome VA score change is ranged from -71 to 52, with the higher VA score change the better visual acuity improvement.
Time Frame: Baseline and 1 Year
Population: All patients who had VA measured at week 52 were included in the analysis. All analyses were performed on the basis of the intention-to-treat principle. The Data and Safety Monitoring Committee recommended that data for all 23 patients at one center be excluded because of serious protocol noncompliance.
Measure: Mean (Standard Deviation); unit: No. of Letters
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 284 | 265 | 285 | 271
No. of Letters | 8.5 (14.1) | 8.0 (15.8) | 6.8 (13.1) | 5.9 (15.7)
Statistical Analysis 1: Comparison: 1-Lucentis Monthly vs 2-Avastin Monthly; The study was designed as a non-inferiority trial among four study groups, with the ability to test for superiority if a treatment was found to be non-inferior. Assuming a standard deviation for changes in visual acuity for 15 letters, we determined that a sample of 277 patients per group (which was increased to 300 to allow for a rate of death or dropout of 8%) would provide a power of 90%; Test type: Non-Inferiority or Equivalence — The non-inferiority limit for the difference between study groups in the mean change in visual acuity at 1 year was 5 letters (i.e., one line on the Early Treatment Diabetic Retinopathy Study [ETDRS] visual-acuity chart); p = 0.16, ANOVA — This p-value is for the test of overall difference among 4 treatment groups. The p-value for pairwise comparison was not performed, because this is a non-inferiority trial; We calcularted of two-sided 99.2% confidence intervals. We used Bonferroni approach to accommodate six pairwise treatment comparisons; Mean Difference (Net) = -0.5, 99.2% CI 2-sided [-3.9 to 2.9], Standard Error of Mean 1.7 — Estimate = Mean VA Change in Avastin Monthly Group - Mean VA Change in Lucentis Monthly Group
Statistical Analysis 2: Comparison: 3-Lucentis as Needed vs 4-Avastin as Needed; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.16, ANOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.8, 99.2% CI 2-sided [-4.1 to 2.4], Standard Error of Mean 1.6 — Estimate = Mean VA Change in Avastin as Needed Group - Mean VA Change in Lucentis as Needed Group
Statistical Analysis 3: Comparison: 1-Lucentis Monthly vs 3-Lucentis as Needed; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.16, ANOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.7, 99.2% CI 2-sided [-4.7 to 1.3], Standard Error of Mean 1.5 — Estimate = Mean VA Change in Lucentis as Needed Group - Mean VA Change in Lucentis Monthly Group
Statistical Analysis 4: Comparison: 2-Avastin Monthly vs 4-Avastin as Needed; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.16, ANOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -2.1, 99.2% CI 2-sided [-5.7 to 1.6], Standard Error of Mean 1.9 — Estimate = Mean VA Change in Avastin as Needed Group - Mean VA Change in Avastin Monthly Group
Statistical Analysis 5: Comparison: 2-Avastin Monthly vs 3-Lucentis as Needed; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.16, ANOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.2, 99.2% CI 2-sided [-4.5 to 2.1], Standard Error of Mean 1.7 — Estimate = Mean VA Change in Lucentis as Needed Group - Mean VA Change in Avastin Monthly Group
Statistical Analysis 6: Comparison: 1-Lucentis Monthly vs 4-Avastin as Needed; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.16, ANOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -2.6, 99.2% CI 2-sided [-5.9 to 0.8], Standard Error of Mean 1.7 — Estimate = Mean VA Change in Avastin as Needed Group - Mean VA Change in Lucentis Monthly Group

3. Secondary Outcome: Visual-acuity Score and Snellen Equivalent (Frequency)
Time Frame: at 1 Year
Measure: Number; unit: Participants
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 284 | 265 | 285 | 271
Participants
  83-97 letters, 20/12-20 | 42 | 45 | 38 | 40
  68-82 letters, 20/25-40 | 149 | 134 | 141 | 127
  53-67 letters, 20/50-80 | 52 | 47 | 66 | 57
  38-52 letters, 20/100-160 | 23 | 21 | 23 | 24
  ≤37 letters, ≤20/200 | 18 | 18 | 17 | 23

4. Secondary Outcome: Visual-acuity Score and Snellen Equivalent (Continuous)
Description: Visual acuity testing was performed with the Electronic Visual Tester (EVA) following the ETDRS protocol. VA score is measured as number of letters read correctly.
  In this study, the outcome VA score is ranged from 0 to 97, with the higher score the better visual acuity.
Time Frame: at 1 Year
Measure: Mean (Standard Deviation); unit: No. of Letters
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 284 | 265 | 285 | 271
No. of Letters | 68.8 (17.7) | 68.4 (18.2) | 68.4 (16.4) | 66.5 (19.0)

5. Secondary Outcome: Number of Treatments
Description: Cumulative over the 1 year of trial
Time Frame: 1 Year
Measure: Mean (Standard Error); unit: Number of Treatments
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 284 | 265 | 285 | 271
Number of Treatments | 11.7 (1.5) | 11.9 (1.2) | 6.9 (3.0) | 7.7 (3.5)

6. Secondary Outcome: Average Cost of Drug/Patient
Time Frame: at 1 Year
Measure: Mean (Standard Deviation); unit: US dollars per patient
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 284 | 265 | 285 | 271
US dollars per patient | 23400 (3000) | 595 (60) | 13800 (6000) | 385 (175)

7. Secondary Outcome: Total Thickness at Fovea
Time Frame: at 1 Year
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 280 | 261 | 281 | 265
μm | 266 (125) | 300 (149) | 294 (139) | 308 (127)

8. Secondary Outcome: Total Thickness Change From Baseline at Fovea
Time Frame: Baseline and 1 Year
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 280 | 260 | 278 | 265
μm | -196 (176) | -164 (181) | -168 (186) | -152 (178)

9. Secondary Outcome: Retinal Thickness Plus Subfoveal-fluid Thickness at Fovea
Time Frame: at 1 Year
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 280 | 261 | 281 | 265
μm | 152 (57) | 172 (81) | 166 (66) | 172 (68)

10. Secondary Outcome: Retinal Thickness Plus Subfoveal-fluid Thickness Change From Baseline at Fovea
Time Frame: Baseline and 1 Year
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 280 | 260 | 278 | 265
μm | -100 (130) | -79 (132) | -81 (134) | -79 (123)

11. Secondary Outcome: Fluid on Optical Coherence Tomography
Time Frame: at 1 Year
Measure: Number; unit: Participants
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 284 | 265 | 285 | 271
Participants
  Absent | 124 | 69 | 68 | 52
  Present | 151 | 188 | 203 | 214
  Data missing | 9 | 8 | 14 | 5

12. Secondary Outcome: Dye Leakage on Angiogram
Time Frame: at 1 Year
Measure: Number; unit: Participants
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 284 | 265 | 285 | 271
Participants
  Absent | 167 | 153 | 133 | 111
  Present | 97 | 100 | 137 | 145
  Data missing | 20 | 12 | 15 | 15

13. Secondary Outcome: Area of Lesion
Time Frame: at 1 Year
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 256 | 243 | 265 | 249
mm^2 | 6.6 (6.8) | 6.5 (6.7) | 7.3 (6.5) | 7.0 (7.5)

14. Secondary Outcome: Area of Lesion Change From Baseline
Time Frame: Baseline and 1 Year
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 250 | 238 | 259 | 241
mm^2 | -0.1 (5.2) | 0.3 (4.9) | 0.6 (6.2) | 1.3 (6.6)

15. Secondary Outcome: Change in Systolic Blood Pressure From Baseline
Time Frame: Baseline and 1 Year
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 239 | 226 | 250 | 232
mm Hg | -2.1 (22.4) | -5.4 (18.2) | -5.2 (20.3) | -4.5 (20.0)

16. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline
Time Frame: Baseline and 1 Year
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Number analyzed (Participants) | 239 | 226 | 250 | 232
mm Hg | -0.9 (11.9) | -1.4 (11.2) | -1.9 (10.2) | -2.1 (10.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at 1 year.
Description: Adverse events were ascertained through monthly questioning of patients by study coordinators who were aware of study-group assignments; events were coded according to the Medical Dictionary for Regulatory Activities (MedDRA) system, version 10. A medical monitor who was unaware of study-group assignments reviewed serious adverse events.
Arm/Group | 1-Lucentis Monthly | 2-Avastin Monthly | 3-Lucentis as Needed | 4-Avastin as Needed
Serious Adverse Events (participants affected / at risk) | 53/301 | 64/286 | 61/298 | 77/300
Other Adverse Events (participants affected / at risk) | 3/301 | 4/286 | 0/298 | 0/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1-Lucentis Monthly (N=301) | 2-Avastin Monthly (N=286) | 3-Lucentis as Needed (N=298) | 4-Avastin as Needed (N=300)
Any other system organ class (General disorders) | 18 | 26 | 16 | 28
Benignor malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5 | 10 | 9
Cardiac disorder (Cardiac disorders) | 10 | 16 | 12 | 13
Death from any cause (General disorders) | 4 | 4 | 5 | 11
Death from vascular causes (Blood and lymphatic system disorders) | 2 | 2 | 2 | 5
Gastrointestinal disorder (Gastrointestinal disorders) | 3 | 6 | 2 | 9
Hypertension (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Infection (Infections and infestations) | 6 | 11 | 12 | 18
Injury or procedural complication (Injury, poisoning and procedural complications) | 7 | 11 | 8 | 9
Nervous system disorder (Nervous system disorders) | 6 | 9 | 12 | 9
Nonfatal myocardial infarction (Cardiac disorders) | 2 | 2 | 3 | 1
Nonfatal stroke (Cardiac disorders) | 3 | 2 | 1 | 2
Surgical or medical procedure (Surgical and medical procedures) | 4 | 6 | 4 | 8
Transient ischemic attack (Cardiac disorders) | 1 | 0 | 2 | 3
Venous thrombotic event (Blood and lymphatic system disorders) | 0 | 4 | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1-Lucentis Monthly (N=301) | 2-Avastin Monthly (N=286) | 3-Lucentis as Needed (N=298) | 4-Avastin as Needed (N=300)
Endophthalmitis (Eye disorders) | 2 | 4 | 0 | 0
Pseudoendophthalmitis (Eye disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Dr. Grunwald reports receiving consulting fees from GlaxoSmithKline; and Dr. Jaffe, consulting fees from Neurotech and SurModics. No other potential conflict of interest relevant to this article was reported.